CLINICAL TRIAL: NCT05012332
Title: A Magnetic Resonance Study to Evaluate the Spread of Local Anesthesia in Healthy Volunteers Receiving an Ultrasound-guided Erector Spinae Plane Block.
Brief Title: Local Anesthesia Spread After an Erector Spinae Plane Block.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Principal Investigator, Marie Sørenstua, Principal investigator, Ostfold Hospital Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 212606
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Regional Anesthesia Morbidity; Postoperative Pain
Keywords: Erector Spinae Plane Block; Magnetic resonance imaging
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: We aim to enroll 10 healthy volunteers. All volunteers receive the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Erector Spinae Plane Block (Other): All volunteers will be given the choice of procedural pain relief in the form of rapifen 0,5-1 mg. All volunteers included will receive an unilateral ESPB at the T7 level with 30 ml of 2,5 mg/ml ropivacaine and a total of 0,3 mmol gadolinium. The intervention will be performed by the PhD candidate connected to the study. The ESPB will be performed under ultrasound guidance, where the needle target is the transverse process of the Th7 vertebra, under the musculus (m.) erector spinae. All volunteers will be tested for cold and pinprick sensation 30 minutes after block completion, and the results plotted on a dermatome map before they undergo an MRI.
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — All volunteers receive an Erector Spinae Plane Block and an MRI.

SUMMARY:
This a single-center prospective spread-evaluation study where the primary objective is to assess the spread of local anesthesia in an ESPB using magnetic resonance imaging (MRI).

The investigators will include 10 healthy volunteers from the hospitals internal website. All volunteers will receive a one-sided Erector Spinae Plane (ESP) block. 30 min after the block sensitivity to cold and pinprick will be assessed before an MRI is performed after 60 min postblock. An radiology specialist will evaluate the MR images pertaining to the spread of the local anesthesia.

DETAILED DESCRIPTION:
Healthy volunteers working at Ostfold Hospital will be recruited by a message put up on the hospitals intranet front page. As participants makes contact, they will receive a mail sent by a study nurse. The mail will include the patient information sheet and a consent form. There will be offered compensation in the form of a gift card of 1000 NOK to cover any travel expenses. Any travel expenses exceeding 1000 NOK will not be covered. If the volunteer fulfills the eligibility criteria and consent is obtained, the study nurse will contact the volunteer per phone or mail to set up an intervention date.

The investigators aim to enroll 10 healthy volunteers and perform the intervention within six months. The planned project end is during December 2022.

All volunteers will be given the choice of procedural pain relief in the form of rapifen 0,5-1 mg. All volunteers included will receive an unilateral ESPB at the T7 level with 30 ml of 2,5 mg/ml ropivacaine and a total of 0,3 mmol gadolinium. The intervention will be performed by the PhD candidate connected to the study. The ESPB will be performed under ultrasound guidance, where the needle target is the transverse process of the Th7 vertebra, under the musculus (m.) erector spinae. All volunteers will be tested for cold and pinprick sensation 30 minutes after block completion, and the results plotted on a dermatome map before they undergo an MRI.

Magnetic resonance imaging study A 3T MRI examination (Magnetom Skyra, Siemens) will be performed 60 minutes after the injection, covering spine levels Th3 to Th12. 3D T1-weighted sequences with fat suppression as well as a T2-weighted sequence will be performed. The distribution pattern of the ropivacaine-gadolinium solution will be evaluated in the following structures: superficial, paravertebral and intercostal musculature, neural foramina and epidural space. All images will be reviewed and analyzed by the same radiologist.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* No comorbidity

Exclusion Criteria:

* Allergy to latex, gadolinium and local anesthesia
* BMI >40
* Severe renal and/or hepatic disease
* Local infection at the site of injection
* Systemic infection
* AV block 2-3
* Inability to understand written or spoken Norwegian
* Inability to cooperate
* Claustrophobia
* Pregnancy - All fertile women will be asked to perform a pregnancy test to ensure that they aren't pregnant before inclusion.
* Metal implants not MRI-compatible

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Local anesthesia spread | 60-120 min
  A 3T MRI examination (Magnetom Skyra, Siemens) will be performed 60 minutes after the injection, covering spine levels Th3 to Th12. 3D T1-weighted sequences with fat suppression as well as a T2-weighted sequence will be performed. The distribution pattern of the ropivacaine-gadolinium solution will be evaluated in the following structures: superficial, paravertebral and intercostal musculature, neural foramina and epidural space.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Soerenstua, MD, Principal Investigator — Sykehuset Ostfold HF
Locations (1):
- Ostfold Hospital Trust, Kalnes, Sarpsborg, Østfold fylke, Norway

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At publication date and for three months.

REFERENCES:
- [Derived] Sorenstua M, Zantalis N, Raeder J, Vamnes JS, Leonardsen AL. Spread of local anesthetics after erector spinae plane block: an MRI study in healthy volunteers. Reg Anesth Pain Med. 2023 Feb;48(2):74-79. doi: 10.1136/rapm-2022-104012. Epub 2022 Nov 9. PMID 36351741